CLINICAL TRIAL: NCT04318015
Title: Chemoprophylaxis With Hydroxychloroquine in Healthcare Personnel in Contact With COVID-19 Patients: A Randomized Controlled Trial (PHYDRA Trial)
Brief Title: Hydroxychloroquine Chemoprophylaxis in Healthcare Personnel in Contact With COVID-19 Patients (PHYDRA Trial)
Acronym: PHYDRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ProfilaxisCOVID
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Severe Acute Respiratory Syndrome
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Triple blinded, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will happen after previous assignment of recruited individual to high-risk or low-risk exposure according to he or her activities. An independent member of the team will randomly assign treatment or placebo following a computer based program. Blinding will end in case elimination criteria are met.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-risk Treatment (Experimental): Hydroxychloroquine 200mg per day for 60 days.
  Interventions: Drug: Hydroxychloroquine
- High-risk Placebo (Placebo Comparator): Placebo tablet per day for 60 days.
  Interventions: Drug: Placebo oral tablet
- Low-risk Treatment (Experimental): Hydroxychloroquine 200mg per day for 60 days
  Interventions: Drug: Hydroxychloroquine
- Low-risk Placebo (Placebo Comparator): Placebo tablet per day for 60 days.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydroxychloroquine — All treatment will be administered orally.
  Other Names: Plaquenil
  Arms: High-risk Treatment; Low-risk Treatment
Drug: Placebo oral tablet — All placebo will be administered orally
  Other Names: Placebo
  Arms: High-risk Placebo; Low-risk Placebo

SUMMARY:
Triple blinded, phase III randomized controlled trial with parallel groups (200mg of hydroxychloroquine per day vs. placebo) aiming to prove hydroxychloroquine's security and efficacy as prophylaxis treatment for healthcare personnel exposed to COVID-19 patients.

DETAILED DESCRIPTION:
Healthcare personnel infection with COVID-19 is a major setback in epidemiological emergencies. Hydroxychloroquine has proven to inhibit coronavirus in-vitro but no data to date has proven in-vivo effects. Nevertheless, hydroxychloroquine is a low cost, limited toxicity and broadly used agent. Since there is currently no treatment for COVID-19 exposure prophylaxis, the investigators will implement a triple blinded, phase III randomized controlled trial with parallel groups (200mg of hydroxychloroquine per day vs. placebo) for 60 days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old upon study start
* Healthcare personnel exposed to patients with COVID-19 respiratory disease: physicians, nurses, chemists, pharmacists, janitors, stretcher-bearer, administrative and respiratory therapists.
* Signed consent for randomization to any study arm.

Exclusion Criteria:

* Known hypersensitivity to hydroxychloroquine manifested as anaphylaxis
* Current treatment to chloroquine or hydroxychloroquine
* Women with last menstruation date farther than a month without negative pregnancy test.
* Women with positive pregnancy test
* Breastfeeding women
* Chronic hepatic disease history (Child-Pugh B or C)
* Chronic renal disease (GFR less or equal to 30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Symptomatic COVID-19 infection rate | From date of randomization until the appearance of symptoms or study completion 60 days after treatment start
  Symptomatic infection rate by COVID-19 defined as cough, dyspnea, fever, myalgia, arthralgias or rhinorrhea along with a positive COVID-19 real-time polymerase chain reaction test.

SECONDARY OUTCOMES:
Symptomatic non-COVID viral infection rate | From date of randomization until the appearance of symptoms or study completion 60 days after treatment start
  Symptomatic infection rate by other non-COVID-19 viral etiologies defined as cough, dyspnea, fever, myalgia, arthralgias or rhinorrhea along with a positive viral real time polymerase chain reaction test.
Days of labor absenteeism | From date of randomization until study completion 60 days after treatment start
  Number of days absent from labor due to COVID-19 symptomatic infection
Rate of labor absenteeism | From date of randomization until study completion 60 days after treatment start
  Absenteeism from labor rate due to COVID-19 symptomatic infection
Rate of severe respiratory COVID-19 disease in healthcare personnel | From date of randomization until the appearance of symptoms or study completion 60 days after treatment start
  Rate of severe respiratory COVID-19 disease in healthcare personnel

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Rojas-Serrano, MD, PhD., Principal Investigator — National Institute of Respiratory Diseases - México; Rogelio Perez-Padilla, MD, Study Director — National Institute of Respiratory Diseases - México; Felipe Jurado-Camacho, MD. MSc, Study Director — National Institute of Respiratory Diseases - México; Ireri Thirion-Romero, MD, MSc, Study Chair — National Institute of Respiratory Diseases - México; Sebastian Rodríguez-Llamazares, MD, MPH, Study Chair — National Institute of Respiratory Diseases - México; Carmen Hernandez Cárdenas, MD, MSc, Study Chair — National Institute of Respiratory Diseases - México; Cristobal Guadarrama-Pérez, MD, Study Chair — National Institute of Respiratory Diseases - México; Alejandra Ramírez-Venegas, MD, MSc, Study Chair — National Institute of Respiratory Diseases - México
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, "Ismael Cosío Villegas", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided